CLINICAL TRIAL: NCT00035061
Title: A Phase 2 Trial of ALIMTA (Pemetrexed) in Locally Advanced or Metastatic Recurrent Transitional Cell Carcinoma of the Urothelium
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Purpose: Treatment
Other Study IDs: 4698; H3E-MC-JMEU; NCT00039260 (obsolete NCT alias)
Record Dates: First submitted 2002-05-02; First posted 2002-05-03 (Estimated); Last update posted 2006-07-19 (Estimated); Status verified 2006-07

CONDITIONS: Urologic Neoplasms; Metastases, Neoplasm
Keywords: Bladder Cancer; Metastatic; Recurrent; Transitional cell carcinoma of the urothelium
MeSH Terms: conditions — Urologic Neoplasms; Neoplasm Metastasis; Urinary Bladder Neoplasms; Recurrence | interventions — Pemetrexed

INTERVENTIONS:
Drug: pemetrexed

SUMMARY:
Patients with bladder cancer will be participating in this study for the treatment of abnormal cells in the bladder that have returned after initial treatment OR have moved to a new site in the body.

ELIGIBILITY:
Inclusion Criteria:

* You must have been diagnosed with bladder cancer that has recurred or moved to a new part of the body.
* You must have at least one tumor that can be physically measured or scanned by x-ray.
* You may not have had previous chemotherapy (drug) treatment OR you have had surgery followed by one chemotherapy treatment at least 4 months ago.

Exclusion Criteria:

* You may not have used an experimental medicine or device within the past month.
* Cancer that has spread to your brain.
* If you are unwilling or unable to take folic acid or vitamin B12 supplements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Los Angeles, California
  - Palo Alto, California
  - Boca Raton, Florida
  - Tampa, Florida
  - Decatur, Illinois
  - Indianapolis, Indiana
  - Lafayette, Indiana
  - Muncie, Indiana
  - South Bend, Indiana
  - Lenexa, Kansas
  - Saint Mathews, Kentucky
  - Boston, Massachusetts
  - Omaha, Nebraska
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Seattle, Washington